CLINICAL TRIAL: NCT00910897
Title: A Phase 3 Study of Velcade (Bortezomib) Dexamethasone (VD) Versus Velcade (Bortezomib) Thalidomide Dexamethasone (VTD) as an Induction Treatment Prior to Autologous Stem Cell Transplantation in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study in Myeloma Patients Newly Diagnosed Treated as an Induction With Velcade-Dex or Velcade (Bortezomib) Thalidomide Dexamethasone (VTD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Intergroupe Francophone du Myelome (Network)
Responsible Party: Principal investigator: HAROUSSEAU Jean-Luc, University Hospital, Nantes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFM 2007-02; Eudract 2007-005204-40
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed; multiple myeloma; induction; Thalidomide
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Velcade-Dexamethasone (Active Comparator)
  Interventions: Drug: Velcade-Dexamethasone
- Velcade-Thalidomide-Dexamethasone (Active Comparator)
  Interventions: Drug: Velcade-Thalidomide-Dexamethasone

INTERVENTIONS:
Drug: Velcade-Dexamethasone
  Arms: Velcade-Dexamethasone
Drug: Velcade-Thalidomide-Dexamethasone
  Arms: Velcade-Thalidomide-Dexamethasone

SUMMARY:
Primary objective:

* Compare the complete remission (CR) rates (i.e., the true CR, with negative immunofixation) achieved with either four courses of VD or four courses of VTD.

Secondary objectives:

* Compare the following parameters following 4 cycles of VD or VTD induction treatment:

  * CR rate+ very good partial remission (VGPR) rate
  * Overall remission rate (CR + VGPR + partial remission (PR) rate)
  * K/l light chain ratio in patients in CR.
  * Safety (quality of the sampled stem cells, extrahaematological and haematological toxicity: specially neurological toxicity, length of hospitalization).
* Compare the CR rate and the CR + VGPR rates after post-induction autologous stem cell transplantation (ASCT).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed symptomatic multiple myeloma (MM) patient
* Aged under 65
* Candidate for ASCT, with measurable levels of paraprotein in the serum (³ 10 g/L) or the urine (³ 200 mg/day)
* Using effective contraceptive methods (for fertile men, women of childbearing potential)
* Provision of informed consent
* No evidence of active infection

Exclusion Criteria:

* Asymptomatic MM
* Non-secretory MM
* Aged 66 years or over
* ECOG performance status over 2 (see Appendix 2)
* Proven amyloidosis
* A personal medical history of cancer (except for basocellular skin cancer or in situ cervical cancer)
* Positive HIV serology
* A personal medical history of severe psychiatric disease
* Severe diabetes contraindicating the use of high-dose dexamethasone
* NCI grade ³ 2 peripheral neuropathy
* Serum clinical chemistry:

  * creatinine level > 300 µmol/L or requiring dialysis
  * bilirubin, transaminases or GamaGT > 3 the upper normal limit (UNL)
* Prior or current systemic therapy for MM, including steroids (except for emergency use of a 4-day block of dexamethasone between the screening phase and randomization)
* Radiation therapy in the 2 weeks preceding randomization
* A personal medical history of allergic reactions to compounds containing boron or mannitol
* Non-controlled or severe cardiovascular disease (including a myocardial infarction in the 6 months prior to recruitment) or NYHA class III or IV renal failure
* Use of any investigational drug in the 30 days preceding randomization
* Pregnant or lactating women; a serum Beta-hCG pregnancy test must be performed during the screening phase for female patients of childbearing potential
* Severe pulmonary troubles (including acute infiltrative pneumopathy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (56):
- Belgium (7):
  - ANVERS Centrumziekenhuis, Antwerp
  - Anvers Uza, Antwerp
  - Bruxelles Erasme, Brussels
  - Bruxelles I Bordet, Brussels
  - BRUXELLES St LUC, Brussels
  - GILLY, Gilly
  - YVOIR MontGodinne, Yvoir
- France (49):
  - Chu Angers, Angers
  - CH Annecy, Annecy
  - Ch Avignon, Avignon
  - CH Bayonne, Bayonne
  - Chu Besancon, Besançon
  - CH BLOIS, Blois
  - Bobigny Avicenne, Bobigny
  - Chu Bordeaux, Bordeaux
  - Chu Brest, Brest
  - Caen M Interne Baclèse, Caen
  - CH Chartres, Chartres
  - Clamart Percy, Clamart
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Ch Colmar, Colmar
  - Chu Dijon, Dijon
  - Ch Dunkerque, Dunkirk
  - Chu Grenoble, Grenoble
  - CH La Roche Sur Yon, La Roche-sur-Yon
  - Le Mans Victor Hugo, Le Mans
  - Chru Lille, Lille
  - Ch Lorient, Lorient
  - CHU Lyon Edouard Herriot, Lyon
  - CHU Lyon Sud Pierre Benite, Lyon
  - Lyon Léon Berard, Lyon
  - Marseille IPC, Marseille
  - CHR Metz Bonsecours, Metz
  - Chu Nancy, Nancy
  - Chu Nantes, Nantes
  - Nantes Catherine De Sienne, Nantes
  - CHU Nice M Interne, Nice
  - CHR Orléans, Orléans
  - Paris Cochin, Paris
  - Paris Hôtel Dieu, Paris
  - Paris Necker, Paris
  - Paris St Antoine, Paris
  - Paris St Louis, Paris
  - CHU Poitiers hemato, Poitiers
  - CHU Reims, Reims
  - CHU Rennes Hemato, Rennes
  - CHU Rennes M interne, Rennes
  - CH Roanne, Roanne
  - Rouen Becquerel, Rouen
  - CH St Brieuc, Saint-Brieuc
  - St ETIENNE, Saint-Etienne
  - CHRU Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - CHU Tours, Tours
  - CH Valence, Valence
  - CH Vannes, Vannes

REFERENCES:
- [Derived] Moreau P, Avet-Loiseau H, Facon T, Attal M, Tiab M, Hulin C, Doyen C, Garderet L, Randriamalala E, Araujo C, Lepeu G, Marit G, Caillot D, Escoffre M, Lioure B, Benboubker L, Pegourie B, Kolb B, Stoppa AM, Fuzibet JG, Decaux O, Dib M, Berthou C, Chaleteix C, Sebban C, Traulle C, Fontan J, Wetterwald M, Lenain P, Mathiot C, Harousseau JL. Bortezomib plus dexamethasone versus reduced-dose bortezomib, thalidomide plus dexamethasone as induction treatment before autologous stem cell transplantation in newly diagnosed multiple myeloma. Blood. 2011 Nov 24;118(22):5752-8; quiz 5982. doi: 10.1182/blood-2011-05-355081. Epub 2011 Aug 17. PMID 21849487